CLINICAL TRIAL: NCT05810662
Title: Randomized Study of Intraoperative Glucose Saline Versus Ringer Lactatein Cancer Pediatric Patients Doing Major Surgeries and Impact on Electrolytes ,Glucose and pH
Brief Title: RL Versus Glucose Saline in Cancer Patient Undergoing Major Surgeries and Its Impact on Electrolytes, GLC & pH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mona Mohammed Atteya, Anesthesia specialist, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AP1907-30106
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Fluid and Electrolyte Imbalance
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ringer lactate (Active Comparator): Ringer's lactate solution, or lactated Ringer's solution, is a type of isotonic, crystalloid fluid further classified as a balanced or buffered solution used for fluid replacement. The contents of Ringer's lactate include sodium, chloride, potassium, calcium, and lactate in the form of sodium lactate, mixed into a solution with an osmolarity of 273 mOsm/L and pH of about 6.5.
  Interventions: Other: Lactated ringer and dextrose 5%
- 5%dextrose in 0.9%saline (Active Comparator): 5% Dextrose and 0.45% Sodium Chloride Injection, USP solution is sterile and nonpyrogenic. It is a large volume parenteral solution containing dextrose and sodium chloride in water for injection intended for intravenous administration.
  Each 100 mL of 5% Dextrose and 0.45% Sodium Chloride Injection, USP contains dextrose, hydrous 5 g and sodium chloride 0.45 g in water for injection. Electrolytes per 1000 mL: sodium (Na+), 77 mEq; chloride (Cl-) 77 mEq. The osmolarity is 406 mOsmol/L (calc.), which is hypertonic. The caloric value is 170 kcal/L.
  The pH is 4.3 (3.5 to 6.5). 5% Dextrose and 0.45% Sodium Chloride Injection, USP contains no bacteriostat, antimicrobial agent or added buffer and is intended only as a single-dose injection.
  Interventions: Other: Lactated ringer and dextrose 5%

INTERVENTIONS:
Other: Lactated ringer and dextrose 5% — Fluid use perioperative

SUMMARY:
To compare two electrolytes maintenance in perioperative period in children undergoing major surgeries on perioperative change in pH,lactate,sodium and glucose level

DETAILED DESCRIPTION:
Patients were randomized into 2 groups ringer lactate versus 5%dextrose in 0.9% saline,using a computer generated random list in blocks of 4 after recruitment the enrolling investigators opened sealed opaque envelopes that concealed group allocation participants ,trial investigators,attending anesthetist providing general anesthesia for the cases and the outcomes were blinded to group allocation

ELIGIBILITY:
Inclusion Criteria:

* 1to 10 years Children undergoing major surgeries ie considered major if any invasive procedure in which extensive resection will be preformed e.g body cavity is opened,organs are removed and normal anatomy is altered abd duration not less than 2 hours or more than 5 hours.

Exclusion Criteria:

* patient guardian refusal

  _ Children with documented endocrine distrubances(DM,inborn error of metabolism,hyperthyroidism)
* age less than one year
* preexisting renal disease,hepatic disease and patien suffering from heart failure.
* preexisting electrolyte imbalance (normal sodium level 135-145)

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-09-04 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
PH and lactate level | In the introperative period
  Three ABG will be collected from the patient. The first at start before any intervention,the second after start of replacement and the third at the end of the operation.

SECONDARY OUTCOMES:
Sodium and glucose level | The intraoperative period
  Three ABGs will be collected.The first at the start of the operation before any surgical intervention,the second after the start of fluid replacement and the last sample at the end of the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Will always be available